CLINICAL TRIAL: NCT04947033
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, MTD or MAD, PK, PD, and Antitumor Activity of TJ210001(a Fully Human C5aR Monoclonal Antibody) in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating TJ210001 in the Treatment of Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ210001STM102
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TJ210001 Injection (Experimental): Single Arm Dose expansion
  Interventions: Drug: TJ210001 Injection

INTERVENTIONS:
Drug: TJ210001 Injection — The test drug TJ210001 will be preset with 5 escalation dose levels: 0.3mg/kg, 1mg/kg, 3mg/kg, 10mg/kg and 15mg/kg, administered once a week.

SUMMARY:
A phase I clinical study evaluating TJ210001 in the treatment of subjects with advanced solid tumors

DETAILED DESCRIPTION:
This study is a phase I clinical study evaluating TJ210001 monotherapy in patients with advanced solid tumors in dose escalation. The overall design of the study is shown in the figure below. The purpose of the TJ210001 single-dose escalation study in subjects with advanced solid tumors is to evaluate the safety and tolerability of monotherapy to determine the MTD (or MAD) and clinically recommended doses of TJ210001 monotherapy.

ELIGIBILITY:
Inclusion Criteria

* Both male and female aged 18 or above;
* ECOG score: 0-1;
* The subjects voluntarily participate in the study, sign the Informed Consent Form, with good compliance, and can cooperate with the follow-up.
* Subjects with advanced malignant solid tumors confirmed by histology or cytology have failed the standard treatment or have no standard treatment protocol or are not suitable for standard treatment at this stage.
* Subjects should have at least one evaluable lesion as defined by RECIST V1.1;
* Subjects who have recovered from the toxicity of previous anti-tumor therapy (CTCAE v5.0) to ≤ Grade 1 or baseline (except for alopecia and neuropathy);
* Expected survival period ≥ 3 months;
* The main organs are functioning normally and the laboratory indicators meet the following standards:

  1. Absolute neutrophil count (ANC) ≥ 1500/μL (≥1.5 ×109/L), and have not received growth factor or colony stimulating factor treatment within 7 days before the start of the study;
  2. Platelets ≥ 75,000/uL (≥100×109/L), and have not received platelet therapy within 14 days before the start of the study;
  3. Hemoglobin ≥8.5g/dL, and have not received blood transfusion treatment in the 14 days before the start of the study (have not received erythropoietin within 3 days before the start of the study);
  4. Adequate renal function and serum creatinine ≤ 1.5×ULN or creatinine clearance ≥ 45 mL/min (calculated by Cockcroft-Gault formula);
  5. Serum total bilirubin ≤ 1.5 × ULN; if diagnosed with Gilbert's disease, serum total bilirubin ≤ 3.0 × ULN; Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3× ULN, or ≤5×ULN for subjects with liver metastasis;
  6. Activated partial thromboplastin time (aPTT) ≤1.5×ULN; International normalized ratio (INR) ≤1.5×ULN (except for anticoagulants with stable doses);
  7. QT interval for QTcF correction and/or QTcB correction of electrocardiogram: male ≤450 ms, female ≤470 ms;
  8. Echocardiography: Left ventricular ejection fraction (LVEF) ≥50%;
* Eligible patients (male and female) with fertility must agree to use reliable contraceptive methods (hormonal or barrier method or abstinence, etc.) with their partners during the study period and at least 90 days after the last administration; Female patients of childbearing age must have a negative blood or urine pregnancy test within 7 days before the first administration of the study drug.

Exclusion Criteria:

* Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before the first administration of the study drug, except for the following items:

  1. Nitrosourea or Mitomycin C has been used within 6 weeks before the first administration of the study drug;
  2. Oral fluorouracil and small molecule targeted drugs are used 2 weeks before the first administration of the study drug or 5 half-lives of the drug (whichever is longer);
  3. Chinese medicine with anti-tumor indications is used within 2 weeks before the first administration of the study drug.
* Have received other unmarketed clinical study drugs or treatments within 4 weeks before the first administration of the study drug;
* Have received major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks before the first administration of the study drug, or the elective surgery will be required during the study period;
* Have received systemic glucocorticoids (prednisone> 10 mg/day or equivalent doses of similar drugs) or other immunosuppressive agents within 14 days before the first administration of the study drug; Except for the following situations: Use topical, eye, intra-articular, intranasal and inhaled glucocorticoid therapy; short-term use of glucocorticoid for preventive treatment (such as prevention of contrast agent allergy)
* Have received immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc. within 14 days before the first administration of study drug;
* Have received the live attenuated vaccine within 4 weeks before the first administration of study drug;
* Have received C5aR inhibitor treatment in the past;
* Those who have previously received allogeneic hematopoietic stem cell transplantation or organ transplantation;
* The adverse reactions of previous anti-tumor treatments have not yet recovered to CTCAE 5.0 grade evaluation ≤ grade 1 (except for the toxicity that the investigator judges to have no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, etc.);
* Patients with central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence indicates that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, and those who are judged by the investigators to be unsuitable for inclusion;
* Those who have an active infection 1 week before the first administration of the study drug and currently require systemic anti-infective treatment;
* Have a history of immunodeficiency, including HIV antibody test positive ;
* Active hepatitis B (HBsAg positive and HBV-DNA > the lower limit of detection of the study center). For subjects who are HBsAg positive but HBV-DNA negative, if the antiviral therapy is needed judged by investigator, the subjects will not be excluded; Hepatitis C virus infection (anti-HCV positive);
* Patients currently suffering from interstitial lung disease;
* Have a history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Have severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia that requires clinical intervention, grade Ⅱ-Ⅲ atrioventricular block;
  2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months before the first administration of study drug;
  3. Patients with the New York Heart Association (NYHA) heart function classification ≥ Grade II;
  4. Have clinically uncontrollable hypertension;
* Patients with active, or have had autoimmune diseases that may have recurrence (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis), except for patients with clinically stable autoimmune thyroid disease;
* Patients who have received immunotherapy and have irAE grade ≥ grade 3;
* Patients who have clinically uncontrollable fluid in the third space and who are judged by the investigator to be unsuitable for enrollment;
* Patients who are known to have alcohol or drug dependence;
* Patients with mental disorders or poor compliance;
* Pregnant or lactating women;
* The subjects who are considered by investigators to have a history of other serious systemic diseases or other reasons are not suitable to participate in this clinical study."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate and Severity of Dose-limiting toxicity （DLT） | up to 28 days after last dose of study drug
Maximum tolerated dose (MTD) | up to 21days following first dose

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No